CLINICAL TRIAL: NCT01316523
Title: Phase II Study of Lenalidomide and Rituximab in Subjects With Previously Untreated Indolent Non Hodgkin's Lymphoma
Brief Title: Lenalidomide and Rituximab in Subjects With Previously Untreated Indolent Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor choice
Sponsor: University of California, Davis (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Joseph Tuscano, Professor, Department of Internal Medicine, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215856; UCDCC#224 (Other: UC Davis); RV_PI_NHL_0488 (Other: Celgene)
Record Dates: First submitted 2011-02-04; First posted 2011-03-16 (Estimated); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: Lenalidomide; Rituximab; untreated indolent Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Rituximab (Experimental): Patients will receive lenalidomide 20 mg daily (oral), on days 1-21 of a 28 day cycle. Rituximab 375 mg/m2 (into the vein) will be administered weekly for 4 doses starting day 15 of cycle 1, to be repeated if patient does not achieve a complete response after cycle 4, on days 1, 8, 15 and 22 of cycle 5.
  Interventions: Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2/wk x 4 weeks, to begin Day 15 of cycle 1. After 4 cycles of therapy if patient does not respond to treatment, the patient will receive a second course of Rituximab.
  Other Names: Rituxan
Drug: Lenalidomide — Lenalidomide will be taken at 20 mg daily, days 1-21 of a 28 day cycle, to be continued until the disease progresses, there are too many side effects, or after twelve cycles if the patient responds to treatment.
  Other Names: Revlimid

SUMMARY:
Lenalidomide has been shown to have single agent activity in indolent Non-Hodgkin's Lymphoma. It is approved for the treatment of multiple myeloma and myelodysplastic syndrome.

Rituximab is effective as a single agent and in combination with chemotherapy for indolent Non-Hodgkin's Lymphoma.

The purpose of this study is to see how well giving lenalidomide together with rituximab works in treating patients with previously untreated indolent Non Hodgkin's Lymphoma.

Lenalidomide will taken at 20 mg daily, days 1-21 of a 28 day cycle, to be continued until the disease progresses, unacceptable side effects or after twelve cycles if the patient is responding well.

Rituximab 375 mg/m2/wk x 4 weeks will begin on Day 15 of cycle 1. After 4 cycles of therapy, if patients respond well to treatment, patients will receive a second course of Rituximab.

Blood samples will be collected to assess how the immune system is functioning.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be informed of the investigative nature of the clinical trial and given written informed consent in accordance with institutional and federal guidelines.
2. Age greater than or equal to 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Previously untreated, histologically confirmed indolent lymphoma including follicle cell lymphoma, WHO classification, grade I or II, and marginal zone lymphoma. Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies. Fine needle aspirates are not acceptable.
5. At least one measurable lesion according to the International Working Group Response criteria for lymphomas. There must be measurable lymphadenopathy to follow with serial exam and/or imaging.
6. Submission of original biopsy for review by local staff hematopathologist.
7. ECOG performance status of 0 -2 at study entry.
8. No major organ dysfunction with laboratory test results within these ranges:

   * Absolute neutrophil count greater than or equal to 1000 /uL
   * Platelet count greater than or equal to 75 x 109/L
   * Total bilirubin less than or equal to 2.0 mg/dL.
   * HIV negative
   * Subjects must have calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance ≥ 30ml/min and < 60ml/min.
9. Life expectancy of greater than 3 months.
10. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
11. Disease free of prior malignancies for greater than or equal to 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
12. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. (patients who are intolerant to aspirin may use low molecular weight heparin).
13. Must be able to swallow lenalidomide capsules.

Exclusion Criteria:

1. Any prior treatment for Non-Hodgkin's Lymphoma.
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
3. Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Known hypersensitivity to thalidomide or rituximab.
7. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
8. Any prior use of lenalidomide.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV
11. Known active hepatitis, type A, B or C.
12. Evidence for CNS metastatic disease
13. Subjects with ≥ Grade 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2024-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Cancer Center, Sacramento, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California

REFERENCES:
- [Derived] Tuscano JM, Dutia M, Chee K, Brunson A, Reed-Pease C, Abedi M, Welborn J, O'Donnell RT. Lenalidomide plus rituximab can produce durable clinical responses in patients with relapsed or refractory, indolent non-Hodgkin lymphoma. Br J Haematol. 2014 May;165(3):375-81. doi: 10.1111/bjh.12755. Epub 2014 Mar 7. PMID 24606326

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide + Rituximab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to Treatment
Description: Responses will be assessed by the Revised Working Group Response Criteria for Malignant Lymphoma. A complete response is the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A partial response is regression of measurable disease and no new sites of disease. Stable disease is failure to attain a complete response/partial response or progressive disease. Response Rate defined as the proportion of patients whose best response was complete response (CR; confirmed or unconfirmed) or partial response (PR).
Time Frame: 4 months
Measure: Number; unit: proportion of patients with CR or PR
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 27
proportion of patients with CR or PR | 0.82

2. Secondary Outcome: Time to Next Treatment.
Description: Time from when the patient started treatment to the time the patient receives next treatment.
Time Frame: Up to about 13 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 27
months | 97.8 [63 to NA] — Upper bound not reached due to study being terminated.

3. Secondary Outcome: Overall Survival
Description: Median overall survival measured as the time from start of treatment to the date of death or the last date the patient was known to be alive.
Time Frame: Up to about 13 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 27
months | NA [NA to NA] — Median OS and 95% Confidence Interval could not be determined because of an insufficient number of participants with events due to the study being prematurely terminated.

4. Secondary Outcome: Number of Patients Experiencing Treatment-related Adverse Events.
Description: Defined as the number of patients experiencing treatment-related adverse events as graded according to the National Cancer Institute Common Toxicity Criteria Version (NCI CTCAE) 4.0.
Time Frame: Up to about 12 years.
Measure: Number; unit: participants
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 30
participants | 28

5. Secondary Outcome: Duration of Response From Start of Therapy
Description: The duration of response is measured from the time measurement criteria are met for complete response/partial response(whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of response is measured from the time measurement criteria are first met for complete response until the first date that recurrent disease is objectively documented.
Time Frame: Up to 14 months.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide + Rituximab
Number analyzed (Participants) | 27
months | 2 [2 to 14]

ADVERSE EVENTS:
Time Frame: About 12 years 9 months
Arm/Group | Lenalidomide + Rituximab
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Rituximab (N=30)
Pancreatitis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Cardiac disorders - Palpitations (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide + Rituximab (N=30)
Anorexia (Metabolism and nutrition disorders) | 5
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 4
Cardiac disorders - Other (Cardiac disorders) | 3
Cataract (Eye disorders) | 2
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 10
Dizziness (Nervous system disorders) | 3
Dry eye (Eye disorders) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 2
Edema face (General disorders) | 2
Edema limbs (General disorders) | 8
Eye disorders - Other (Eye disorders) | 3
Fall (Injury, poisoning and procedural complications) | 4
Fatigue (General disorders) | 14
Fever (General disorders) | 6
Flu like symptoms (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Gait disturbance (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 6
General disorders and administration site conditions - Other (General disorders) | 2
Generalized muscle weakness (General disorders) | 3
Headache (Nervous system disorders) | 6
Hematoma (Vascular disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Hot flashes (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Infections and infestations - Other (Infections and infestations) | 5
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2
Insomnia (Psychiatric disorders) | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 2
Lung infection (Infections and infestations) | 3
Lymphocyte count decreased (Investigations) | 7
Malaise (General disorders) | 2
Memory impairment (Nervous system disorders) | 2
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Nervous system disorders - Other (Nervous system disorders) | 6
Neutrophil count decreased (Investigations) | 4
Non-cardiac chest pain (General disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5
Platelet count decreased (Investigations) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3
Sinusitis (Infections and infestations) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 10
Skin infection (Skin and subcutaneous tissue disorders) | 3
Syncope (Nervous system disorders) | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Upper respiratory infection (Infections and infestations) | 10
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract infection (Renal and urinary disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 2
Vertigo (Ear and labyrinth disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
White blood cell decreased (Investigations) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT01316523/Prot_SAP_000.pdf